CLINICAL TRIAL: NCT02045927
Title: BIS-Guided Sedation Monitoring: A Prospective Randomized Study
Brief Title: BIS-Guided Sedation Monitoring
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: study staff change
Sponsor: Englewood Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-13-519
Record Dates: First submitted 2014-01-22; First posted 2014-01-27 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Patients Who Are Mechanically Ventilated and Sedated
Keywords: sedation; BIS; monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intevention Group (Active Comparator): sedation monitoring with RASS score plus sedation monitoring with BIS-Guided monitoring
  Interventions: Other: sedation monitoring with RASS score; Other: sedation monitoring with BIS-Guided monitoring
- Control Group (Other): sedation monitoring with RASS score
  Interventions: Other: sedation monitoring with RASS score

INTERVENTIONS:
Other: sedation monitoring with RASS score
Other: sedation monitoring with BIS-Guided monitoring
  Arms: Intevention Group

SUMMARY:
This study looks to assess whether monitoring sedation status in mechanically-ventilated Medical Surgical Intensive Care Unit (MSICU) patients using Bispectral index (BIS) monitor-augmented sedation monitoring as opposed to Richmond Agitation Sedation Scale (RASS) score is associated with decreased duration of mechanical ventilation.

Investigators hypothesize that using BIS monitors to help monitor depth of sedation in mechanically ventilated ICU patient will result in a decreased duration of mechanical ventilation when compared to solely utilizing clinical sedation scales such as RASS.

DETAILED DESCRIPTION:
Participants will be randomized into two groups, the intervention group will receive sedation monitoring with BIS monitoring plus RASS. The control group will receive sedation monitoring with RASS score only. Randomization will be accomplished through online randomization software.

For randomization purposes, the intervention group will be labeled as the "A" group. The control group will labeled as the "B" group. In the BIS-augmented group, sedation requirement will be titrated according to an average of BIS reading in the 5 minute period prior to assessment with a goal of maintaining a value of (60-70) in addition to a RASS score goal of (-1 to -2), provided no noxious stimulation such as endotracheal suctioning and/or wound dressing has occurred for at least 30 minutes, BIS values have been stable for at least 5 minutes, signal quality index (>80%), minimal EMG interference (<50%), patient is not shivering, and patient does not have warmer or other devices that may produce an electric current on their body or nearby. In the RASS group, sedation requirements will be titrated to maintain a RASS score of (-1 to -2), will be assessed via the nurse taking care of the patient provided no noxious stimulation has occurred for at least 30 minutes prior to assessment.

Both groups will have sedation assessment at least every 6 hours during a 12 hour shift and as needed as per ICU RN and/or physician. Nurses will be free to exercise their judgment if they deem that their patients require more or less sedation that is inconsistent with patient's BIS or RASS score, they will, however, be required to provide a rationale for their judgment and record such events on a special form created for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age.
* Patients expected to be mechanically ventilated and sedated with continuous intravenous infusions of Propofol or Midazolam and fentanyl for >= 24 hours within 12 hours of screening.

Exclusion Criteria:

* Patients with Seizure disorders acute neurological injury, severe dementia or anoxic brain injury.
* Patients with tracheostomies.
* Patients requiring neuromuscular blocking agents (NMBA).
* Patients transferred from another ICU while mechanically ventilated.
* Patients with cardiac pacemakers.
* Peri-cardiac arrest patients.
* Patients with induced hypothermia.
* Pregnant patients.
* Patients with no known Legally Authorized Representative (LAR).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
duration of mechanical ventilation | from enrollment to extubation, an expected average of 4 days

SECONDARY OUTCOMES:
total sedation medication dose | from enrollment until extubation, an expected average of 4 days
undersedation | from enrollment to extubation, an expected average of 4 days
  measured by self-initiated medical support device removal, time in hours spent in physical restraints, or ventilator asynchrony

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Gianatiempo, MD, Principal Investigator — Englewood Hospital and Medical Center
Locations (1):
- Englewood Hospital and Medical Center, Englewood, New Jersey, United States